CLINICAL TRIAL: NCT01473706
Title: Mini Nutritional Assessment: Consumer Validation
Brief Title: Validation of a Nutrition Screening Tool
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 11.01.US.HCN
Record Dates: First submitted 2011-11-10; First posted 2011-11-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Malnutrition
Keywords: Malnutrition; Nutrition status; Elderly; Nutrition screening
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Consumers: Adults aged ≥ 65 years; Employed part-time, unemployed, retired, full-time or a homemaker; English speaking
  Interventions: Other: Consumer Mini Nutritional Assessment
- Caregivers of Consumers: Family, relative, friend, professional caregiver of an individual age ≥ 65 years; Lives with individual aged ≥ 65 years OR Visits individual aged ≥ 65 years five or more days a week; Makes decisions or has strong influence on the individual aged ≥ 65 years' diet and medical needs; English speaking
  Interventions: Other: Consumer Mini Nutritional Assessment

INTERVENTIONS:
Other: Consumer Mini Nutritional Assessment — A 11 question, self administered nutrition screening tool. The consumer and their caregiver will complete the consumer version of the Mini Nutritional Assessment. A healthcare professional will then meet with the consumer and complete a nutrition screening with utilizing a validated nutrition screening tool.

SUMMARY:
The purpose of this study is to compare the accuracy of a new consumer nutrition screening tool to an established and validated nutrition screening tool currently completed by healthcare practitioners.

DETAILED DESCRIPTION:
The main objective of the study is to determine the accuracy of the self-administered consumer Mini Nutritional Assessment by comparing the level of agreement in the categorization of nutritional status between the self-administered Mini Nutritional Assessment and a validated nutrition screening tool in a population aged 65 and older.

ELIGIBILITY:
Inclusion Criteria:

- Consumer

* Age ≥ 65 years
* Employed part-time, unemployed, retired, full-time homemaker
* English speaking

  - Caregiver of Consumer
* Family, relative, friend, professional caregiver of an individual age ≥ 65 years
* Lives with individual aged ≥ 65 years OR Visits individual aged ≥ 65 years five or more days a week

  * Makes decisions or has strong influence on the individual aged ≥ 65 years' diet and medical needs.
* English speaking

Exclusion Criteria:

- Consumer

-- Full time employment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Consumers aged 65 or older with or without their caregiver
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity and the specificity (in percent) of the consumer version of the Mini Nutritional Assessment versus a validated nutrition screening tool | Within a one hour visit

SECONDARY OUTCOMES:
Ability of the consumer version of the Mini Nutritional Assessment to predict the accuracy of the nutrition status classifications (normal nutritional status, at risk of malnutrition & malnourished) | Within a one hour visit

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Lehrhaupt, Principal Investigator — Kantar Health
Locations (1):
- Kantar Health, New York, New York, United States